CLINICAL TRIAL: NCT06013787
Title: "Nuestras Historias": Evaluating the Impact of Community-Created Digital Stories on Pre- and Perinatal Health Motivation in the Peruvian Amazon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0000065203
Record Dates: First submitted 2018-10-17; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2018-08

CONDITIONS: Health Knowledge, Attitudes, Practice; Maternal Behavior
Keywords: Community-based participatory research; Digital storytelling; Maternal child health; Community health workers; Behavior change communication; Low-resource settings
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Cluster-matched randomized trial, by community, with 5 intervention communities and 5 control communities
Masking Description: Participants were made aware through the informed consent that 1/2 of the communities would be receiving a video intervention. Care providers (community health workers who delivered the video intervention) were trained in it so were not blinded. Outcomes assessor was investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the communities randomized into the intervention arm, the pregnant women who enrolled in the study received a month long prenatal health education intervention called "Nuestras Historias", a digital story curriculum. This video-based curriculum was delivered by by community health workers during their normal home visits and group visits.
  Interventions: Behavioral: "Nuestras Historias"
- Control Group (No Intervention): In the communities randomized to the control arm, the pregnant women who enrolled in study had normal visits and group visits with community health workers and received standard prenatal health education, but with no video intervention.

INTERVENTIONS:
Behavioral: "Nuestras Historias" — "Nuestras Historias" is a digital story curriculum that is displayed on a small solar-powered tablet. The curriculum is a collection of 7 digital stories used to discuss health issues during pregnancy that the community identified as important. The digital stories are short videos that combine local photos and local voices sharing real-life narratives about experiences during pregnancy. The videos were made in collaboration with community health workers and local mothers.
  Other Names: A Digital Story Curriculum on Prenatal Health
  Arms: Intervention Group

SUMMARY:
"Nuestras Historias" curriculum is a tablet-based digital story curriculum that was created through community-based participatory methods. It uses narrative videos to teach about local prenatal health issues in the Parinari District of Peru. This study aims to assess the impact of "Nuestras Historias" on pregnant women and their partners by measuring participants' changes in prenatal health knowledge, attitudes and behavioral intentions for pregnancy and birth after exposure to the curriculum. The study uses a cluster-randomized design, in which communities were match-paired and then randomized for pregnant women/partners to receive the "Nuestras Historias" curriculum vs. standard prenatal health teaching, delivered by local community health workers.

DETAILED DESCRIPTION:
Background and Study Setting:

Parinari is a district in the Loreto region that has 30 communities with approximately 7264 people. The communities are very dispersed and only accessible by river. Inhabitants of this district do not have access to running water, electricity or sanitation and the majority live in poverty. Our study takes place in the 13 communities of Parinari where the Mama River project operated. Mama River selects community health workers (CHWs) who are able to use smartphones in these communities and trains them on the use of smartphones to collect information of new pregnancies, deliveries, alarms signs or deaths of pregnant women or newborns. CHWs then send this information via mobile phone to local health care providers. CHWs are also all trained in the delivery of verbal MCH educational messages to pregnant women, and perform home visits and group visits throughout pregnancies.

Methods:

Twelve communities (6 intervention, 6 control) were recruited and after a final evaluation we excluded two communities, as one had no pregnant women at time of study initiation. The remaining communities were divided into 5 pairs, where the two within the pair were similar in terms of overall population, distance from a health center, and number of pregnant women. One community in each pair was randomly assigned to the intervention group received the Mama River programming along with the digital story curriculum, and the other community to the control group, which received only the standard existing program with no digital stories.

The community agents in the five communities selected for the intervention received training on how to use and show the digital stories on solar-powered tablets.

During the recruitment phase, all pregnant women identified by Mama River were recruited into the trial, with an effort to also recruit their partners. All trial participants signed an informed consent prior to participating, and then completed the pre-intervention survey instrument that measured prenatal health knowledge, attitudes, and behavioral intentions for pregnancy and birth.

Then, in the intervention communities, the participants received home visits and attended group meetings with the community agent in which the digital story curriculum was shown and discussed. In the control communities, participants also received home visits and attended group meetings, but the community agents carried on their standard of practice without the digital stories.

One month after completing the pre-survey, participants completed a post-survey. Those in the intervention group had a slightly longer survey including a short quantitative questions regarding their reactions to the digital stories.

ELIGIBILITY:
Inclusion Criteria:

* All female participants had to be confirmed pregnancies, living permanently within the selected communities of the Parinari District, and age 18 or older
* All male participants had to be partners of women who were confirmed to be pregnant, living permanently within the selected communities of the Parinari District, and age 18 or older

Exclusion Criteria:

* Participants were excluded if not pregnant, if not living in the correct communities or likely to travel away within the study time frame, or if did not consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2016-05-21 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Prenatal Health Knowledge Change | Pre and post one month intervention
  Change in understanding of basic prenatal health information covered in curriculum, measured using our study's survey tool, which included knowledge questions from several validated studies and from the Peruvian government's manual for community health agents, total possible score of 45
Prenatal Health Attitude Change | Pre and post one month intervention
  Change in attitudes towards local issues associated with pregnancy, measured via our study's survey tool with tailored questions to topics that are covered in the curriculum (adolescent pregnancy, domestic violence), and a previously validated measure on locus of control, total possible score of 8
Change in Behavioral Intentions | Pre and post one month intervention
  Change in reported behavioral intentions for practices during pregnancy and at time of birth, measure via our study's survey tool, with a series of questions about the expected birth plan based on the Peruvian government's community agent guide and some video-specific questions, total possible score of 6

CONTACTS AND LOCATIONS:
Overall Officials: Neha Limaye, MD, Principal Investigator — Fellow at UPCH and UW
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: Undecided
At present, all data is securely stored. If study is published, de-identified data will be made available via a secure sharing method.